CLINICAL TRIAL: NCT03402893
Title: The Use of Onexton in Moderate Acne Vulgaris for Patients With Skin of Color
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Principal Investigator, L.H. Kircik, M.D., Medical Director, Derm Research, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONX-1701
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2019-02-19 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Acne Vulgaris; Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm Onexton gel application (Experimental): Onexton gel will be supplied to all subjects and applied once daily to the face
  Interventions: Drug: ONEXTON Topical Gel

INTERVENTIONS:
Drug: ONEXTON Topical Gel — Onexton gel applied once daily to face

SUMMARY:
This is a single-center, open label pilot study. The study is comprised of 5 study visits; Screening, Baseline, and Weeks 4, 8, and 16. All subjects will receive Onexton at Baseline and be instructed to apply the gel once daily to the face. The investigators will evaluate Investigator Global Assessment of acne (IGA), total lesion count, inflammatory lesion count, non-inflammatory lesion count, Investigator Global Assessment of Post-Inflammatory Hyperpigmentation and distribution of Post-Inflammatory Hyperpigmentation, adverse events and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

i. Outpatient, subjects of skin of color, age 12 or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study;

A female is considered of childbearing potential unless she is:

* postmenopausal for at least 12 months prior to study drug administration
* without a uterus and/or both ovaries; or
* has been surgically sterile for at least 6 months prior to study drug administration

Reliable methods of contraception are:

* intrauterine device in use ≥ 90 days prior to study drug administration;
* barrier methods plus spermicide in use at least 14 days prior to study drug administration; or
* vasectomized partner

[Exception: Female subjects of childbearing potential who are not sexually active will not be required to practice a reliable method of contraception. These subjects may be enrolled at the Investigator's discretion if they are counseled to remain sexually inactive during the study and understand the possible risks in getting pregnant during the study.]

ii. Facial acne vulgaris in patients with skin of color (Fitzpatrick Type V & VI Supplement VI) characterized by the following:

* IGA Score for acne vulgaris 3
* IGA Score for PIH 3

iii. Able to understand and comply with the requirements of the study and sign Informed Consent /HIPAA Authorization forms

Exclusion Criteria:

i. Female subjects who are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control

ii. Allergy/sensitivity to any component of the test treatment

iii. IGA score for acne of 2 (mild) or 4 (severe)

iv. IGA score for Post Inflammatory Hyperpigmentation of 2 (mild) or 4 (severe)

v. Subjects who have not complied with the proper wash-out periods for prohibited medications (Supplement I).

vi. Medical condition that, in the opinion of the Investigator, contraindicates the subject's participation in the clinical study

vii. Skin disease/disorder that might interfere with the diagnosis or evaluation of acne vulgaris

viii. Evidence of recent alcohol or drug abuse

ix. History of poor cooperation, non-compliance with medical treatment, or unreliability

x. Exposure to an investigational study drug within 30 days of the Baseline Visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant signed consent but failed screening
Groups:
- Onexton Gel Application: Onexton gel (clindamycin phosphate 1.2%/benzoyl peroxide 3.75%) will be supplied to all subjects and applied once daily to the face
  ONEXTON Topical Gel: Onexton gel applied once daily to face
Period: Overall Study
Arm/Group | Onexton Gel Application
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Facial Investigator Global Assessment of Disease Severity [Count of Participants; unit: Participants] — This assessment measures the severity of acne. The minimum value is 0/Absent and the maximum value is 5/severe. The data is reported as the percentage of patients who fall into each category at each time point.
  Participants
    Moderate | 20
    Clear | 0
    Almost Clear | 0
    Mild | 0
    Severe | 0
Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesion] | 14 (5)
Non-Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesion] | 15 (4)
Post Inflammatory Hyperpigmentation Distribution [Count of Participants; unit: Participants] — Each category describes the extent of facial distribution of post-inflammatory hyperpigmentation
  Participants
    1-10% | 2
    11-20% | 3
    21-30% | 6
    31-40% | 4
    41-50% | 3
    over 50% | 2
Total Lesion Count [Mean (Standard Deviation); unit: lesion] | 29 (4)
Investigator Global Assessment of Severity of Facial Post Inflammatory Hyperpigmentation [Count of Participants; unit: Participants] — This assessment measures the severity of facial post-inflammatory hyperpigmentation. The minimum value is None and the maximum is Moderately Severe. The results are reported as the number of subjects falling under each category and the corresponding percentage of total participants falling under each category.
  Participants
    None | 0
    Slight | 0
    Mild | 0
    Moderate | 20
    Moderately Severe | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment Scale for Severity of Facial Acne
Description: Percent of subjects achieving clear or almost clear on Investigator's Global Assessment (IGA) scale for facial acne; the IGA scale for acne reflects the Investigator's assessment of the severity of a subject's acne on a scale from 0 to 5 with 0 = Clear Skin, 1 = Almost Clear, 2 = Mild, 3 = Moderate severity, 4 = Severe, 5 = Very Severe Each of these gradations is based upon a lesion count by the Investigator.
Time Frame: Week 4, Week 8, Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
Participants
  week 4: clear | 0
  week 4: almost clear | 0
  week 4: mild | 11
  week 4: moderate | 9
  week 4: severe | 0
  week 8: clear | 0
  week 8: almost clear | 6
  week 8: mild | 12
  week 8: moderate | 2
  week 8: severe | 0
  week 16: clear | 1
  week 16: almost clear | 13
  week 16: mild | 6
  week 16: moderate | 0
  week 16: severe | 0

2. Primary Outcome: Investigator Global Assessment Scale for Severity of Post Inflammatory Hyperpigmentation
Description: Percent of subjects achieving clear or almost clear on Investigator's Global Assessment (IGA) scale for severity of post inflammatory hyperpigmentation; the IGA scale of post-inflammatory hyperpigmentation reflects the Investigator's assessment of the severity of a subject's hyperpigmentation on a scale from 0 to 6 with 0 = None, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = moderately Severe, 5 = Severe, 6 = Very severe Each of these gradations is based upon the investigator's impression
Time Frame: Week 4, Week 8, Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
Participants
  week 4: none | 0
  week 4: slight | 2
  week 4: mild | 17
  week 4: moderate | 1
  week 4: moderately severe | 0
  week 8: none | 0
  week 8: slight | 2
  week 8: mild | 15
  week 8: moderate | 2
  week 8: moderately severe | 1
  week 16: none | 0
  week 16: slight | 8
  week 16: mild | 11
  week 16: moderate | 1
  week 16: moderately severe | 0

3. Secondary Outcome: Percent Change in Inflammatory Lesions
Description: The Investigator will count the number of facial (from hairline to mandibular line) inflammatory acne lesions at each study visit. Inflammatory lesions include papules, pustules and nodules.
Time Frame: Week 4, Week 8, Week 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
percent change
  Week 4 | -35 (17)
  Week 8 | -55 (22)
  Week 16 | -76 (14)

4. Secondary Outcome: Percent Change in Non-inflammatory Lesion Count
Description: The Investigator will count the number of facial non-inflammatory acne lesions at each study visit. these include open and closed comedones.
Time Frame: Week 4, Week 8, Week 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
percent change
  week 4 | -21 (22)
  week 8 | -41 (33)
  week 16 | -62 (32)

5. Secondary Outcome: Percent Change in Total Lesion Count
Description: The Investigator will count the number of facial inflammatory and non-inflammatory acne lesions at each study visit. These include papules, pustules, nodules, and open and closed comedones.
Time Frame: week 4, Week 8, Week 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Onexton Gel Application
Number analyzed (Participants) | 20
percent change
  week 4 | -29 (17)
  week 8 | -51 (21)
  week 16 | -71 (13)

6. Secondary Outcome: Post-Inflammatory Hyperpigmentation (PIH) Distribution
Description: This measure as assessed by the Investigator seeks to quantify the extent to which post-inflammatory hyperpigmentation is distributed across the face, wherein 0= No PIH, 1=1-10% of the face affected, 2=11-20%, 3=21-30%, 4=31-40%, 5=41-50%, and 6=More than 50% of the face. Lower numbers reflect less severe disease.
Time Frame: baseline, Week 4, week 8, week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Onexton Gel Application
Number analyzed (Participants) | 20
Participants
  Baseline: 0 | 0
  Baseline: 1 | 2
  Baseline: 2 | 3
  Baseline: 3 | 6
  Baseline: 4 | 4
  Baseline: 5 | 3
  Baseline: 6 | 2
  week 4: 0 | 0
  week 4: 1 | 2
  week 4: 2 | 3
  week 4: 3 | 7
  week 4: 4 | 3
  week 4: 5 | 3
  week 4: 6 | 2
  week 8: 0 | 0
  week 8: 1 | 2
  week 8: 2 | 4
  week 8: 3 | 8
  week 8: 4 | 3
  week 8: 5 | 2
  week 8: 6 | 1
  week 16: 0 | 0
  week 16: 1 | 5
  week 16: 2 | 5
  week 16: 3 | 5
  week 16: 4 | 4
  week 16: 5 | 1
  week 16: 6 | 0

ADVERSE EVENTS:
Time Frame: screening to week 16
Arm/Group | Onexton Gel Application
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onexton Gel Application (N=20)
intermittent mid back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
group A beta hemolytic strep pharyngitis (Infections and infestations) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cellulitis right knee (Infections and infestations) | 1 (1)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pharyngitis (Skin and subcutaneous tissue disorders) | 2 (2)
unexpected menses (Reproductive system and breast disorders) | 1 (1)
facial tattoo tightening (Skin and subcutaneous tissue disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chest soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
serous otitis media (Ear and labyrinth disorders) | 1 (1)
bacterial vaginosis (Reproductive system and breast disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
maxillary fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT03402893/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT03402893/Prot_SAP_001.pdf